CLINICAL TRIAL: NCT03976557
Title: Implementation and Evaluation of BIP CVC in Access Center at Danderyd Hospital, Stockholm, Sweden. Study Protocol
Brief Title: BIP CVC in Access Center at Danderyd Hospital, Stockholm, Sweden
Acronym: IMPROWE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Corona/Covid19 pandemic
Sponsor: Bactiguard AB (Industry)
Collaborators: Danderyd Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PL-13732
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Vascular Access Complication; Catheter-Related Infections; Catheter Thrombosis; Catheter Blockage; Catheter Complications; Catheter Site Discomfort; Catheter Bacteraemia
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Intervention Model Description: Pilot, randomized, open label, controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIP CVC (Experimental): Polyurethane CVC with noble metal coating
  Interventions: Device: BIP CVC
- Standard CVC (Active Comparator): Standard CVC made of polyurethane
  Interventions: Device: Standard CVC

INTERVENTIONS:
Device: BIP CVC — Central venous access with noble metal coated CVC
  Other Names: Noble metal coated CVC
  Arms: BIP CVC
Device: Standard CVC — Central venous access with standard uncoated CVC
  Other Names: Uncoated CVC
  Arms: Standard CVC

SUMMARY:
Primary objective of the study is to establish the incidence of all any catheter related complications in BIP CVC and standard CVC groups in patients requiring CVC.

(CVC - Central Venous Catheter; BIP - Bactiguard Infection Protection)

DETAILED DESCRIPTION:
Catheter related complications include CRBSI, CRI, Local CVC infection, need to exchange of CVC due to suspected CRI/CRBSI or thrombosis, stop / slower flow in any CVC lumen, local thrombosis, device malfunctions / technical catheter problems, device related adverse events.

(CRBSI - Catheter Related Blood Stream Infection; CRI - Catheter Related Infection)

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the Access Center at Danderyd who need an elective CVC (surgery, infection, nutrition, medication…)
2. Fully recognize and understand patient information
3. Signed informed consent

Exclusion Criteria:

1. If CVC present prior to inclusion in the study and no intention to change the present CVC over guidewire
2. Age < 18 years
3. Pregnant women
4. Known allergy to gold, silver and palladium
5. Participation in other clinical studies which may interfere with this study as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Number of patients with catheter related complications | From CVC insertion until CVC withdrawal
  Patients having any complication specified as secondary endpoints

SECONDARY OUTCOMES:
Number of patients with CRBSI | From CVC insertion until CVC withdrawal
  CRBSI - Catheter Related Blood Stream Infections
Number of patients with CRI | From CVC insertion until CVC withdrawal
  CRI - Catheter Related Infections
Number of patients with local CVC infections | From CVC insertion until CVC withdrawal
  Skin infection at the insertion site
Number of CVC exchanges per patient due to suspected infection or thrombosis | From CVC insertion until CVC withdrawal
  Reported as incidence
Number of patients with stop or slower flow in any CVC lumen | From CVC insertion until CVC withdrawal
  Stop or slower flow or need of high pressure during blood sample withdrawal and/or injection of solution
Number of patients with local thrombosis | From CVC insertion until CVC withdrawal
  Local thrombosis - thrombosis in the insertion vein
Number of patients with device malfunctions | From CVC insertion until CVC withdrawal
  Any device malfunction or technical problems during insertion, withdrawal or use
Number of patients with antibiotics and antithrombotics drug use | From CVC insertion until CVC withdrawal
  including the reason of use and dose / number of days
Number of patients with adverse events | From CVC insertion until CVC withdrawal
  including casuality assessment to the CVC use; both serious and non-serious

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jakobsson, Prof, Principal Investigator — Danderyd Hospital
Locations (1):
- Danderyd Sjukhus, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No